CLINICAL TRIAL: NCT04349813
Title: Analysis of Perioperative Pediatric Blood Transfusion Therapy
Brief Title: Perioperative Pediatric Blood Transfusion Therapy
Status: Completed | Type: Observational
Sponsor: Johann Wolfgang Goethe University Hospital (Other)
Responsible Party: Principal Investigator, Dr. Florian Piekarski, Principal Investigator, Johann Wolfgang Goethe University Hospital
Other Study IDs: KGU_FP_2020_CA11
Record Dates: First submitted 2020-04-09; First posted 2020-04-16 (Actual); Last update posted 2020-08-24 (Actual); Status verified 2020-08

CONDITIONS: Transfusion
Keywords: Transfusion, Pediatric, Patient Blood Management

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The present retrospective study analyses perioperative haemotherapy in children and adolescents at the University Hospital Frankfurt.

DETAILED DESCRIPTION:
In the center of the analyses are the perioperative consumption of transfused red cell concentrates, platelet concentrates and frozen fresh plasma in children and adolescents. The distribution by subject area is also examined, demographic distribution and indicators on transfusion. With the introduction of the Patient Blood Management for adults at the University Hospital in 2013 have become potentially also result in changes in transfusion practice in children, which should also be investigated.

ELIGIBILITY:
Inclusion Criteria:

* Children and adolescents <18 years
* Hospital admission
* Operation

Exclusion Criteria:

- none

Max Age: 17 Years | Sex: All
Age Groups: Child
Gender Based: Yes
Study Population: Children undergoing surgery
Sampling Method: Probability Sample
Enrollment: 14248 (Actual)
Dates: Start 2020-04-15 (Actual); Primary Completion 2020-08-01 (Actual); Study Completion 2020-08-01 (Actual)

PRIMARY OUTCOMES:
Transfused red cell concentrates | 01.01.2010 - 31.12.2019
  Quantity of transfused red cell concentrates
Platelet concentrates transfused | 01.01.2010 - 31.12.2019
  Quantity of Platelet concentrates transfused

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anaesthesiology, Intensive Care Medicine and Pain Therapy, University Hospital Frankfurt, Goethe University, Frankfurt, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: No